CLINICAL TRIAL: NCT00238472
Title: A Pilot Study to Evaluate the Effects of Nateglinide vs. Glibenclamide on Renal Hemodynamics and Albumin Excretion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDJN608AIT05
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes; nateglinide
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nateglinide

INTERVENTIONS:
Drug: nateglinide

SUMMARY:
This study is not being conducted in the United States. The purpose of the study is to evaluate the effects of nateglinide compared to glibenclamide on renal hemodynamics and albumin excretion.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes diagnosed at least 1 year before inclusion
* Blood glucose criteria must be met
* Microalbuminuria criteria must be met

Exclusion Criteria:

* Pregnant or nursing females or females of childbearing potential not using a medically approved birth control method
* Blood glucose criteria outside the specified range
* Microalbuminuria criteria outside the specified range
* Serious cardiovascular events within the past 6 months
* Other protocol-defined exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-05; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial glomerular filtration rate at 12 weeks

SECONDARY OUTCOMES:
Change from baseline in fasting morning glomerular filtration rate at 12 weeks
Change from baseline in postprandial renal plasma flow at 12 weeks
Change from baseline in fasting morning renal plasma flow at 12 weeks
Change from baseline in adjusted 2-hour postprandial glucose at 12 weeks
Change in insulin AUC (0-240 minutes) at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals